CLINICAL TRIAL: NCT04000269
Title: Pilot Study Using Targeted High Definition Transcranial Direct Current Stimulation to Promote Upper Extremity Motor Function in Patients With Subacute Middle Cerebral Artery (MCA) Stroke
Brief Title: HD-tDCs to Improve Upper Extremity Function in Patients With Acute Middle Cerebral Artery Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive IRB approval
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: None at this time
Record Dates: First submitted 2019-04-01; First posted 2019-06-27 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Middle Cerebral Artery Stroke
MeSH Terms: conditions — Infarction, Middle Cerebral Artery

STUDY DESIGN:
Intervention Model Description: Pilot prospective double blinded randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Treatment with 'Soterix MxN Neuromodulation device (high definition transcranial direct current stimulator) using HD-Targets for optimal neural targeting will be provided to participants and will include 20 minutes of stimulation coupled with conventional OT treatment during and after the intervention. There will be a total of 10 sessions over about a 2 week period.
  Interventions: Device: Soterix MxN Neuromodulation device
- Sham group (Sham Comparator): Sham stimulation will consist of using the devices auto-sham feature. The exact same setup/device will be used during both groups. This is considered a control for the experiment. Both groups will receive similar physical occupational and speech therapy
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Soterix MxN Neuromodulation device — Up to 2 mA stimulation to primary motor cortex for 10 sessions at 20min per session
  Arms: Treatment Group
Device: Sham Stimulation — Uses slight stimulation initially then turns of and provides no stimulation after a few seconds.
  Arms: Sham group

SUMMARY:
To determine if using targeted high definition transcranial direct current stimulation can improve upper extremity motor function in patients with subacute middle cerebral artery (MCA) stroke.

DETAILED DESCRIPTION:
Current research suggests there may be potential benefit using high definition transcranial direct current stimulation in patients with upper extremity hemiparesis secondary to an ischemic stroke. The intervention has effects on the damaged neurons within the person's brain after stroke possibly amplifying the body's own healing process. These data are compelling but not always statistically significant, which could be due to several reasons. One is the lack of a definitive protocol involving timing of the intervention relative to therapy, lead placement, an unclear dose-response relationship, and variable conductance of tissue and skull thickness. Hummel et al (2008) suggested that stimulation during or before intensive therapy yielded improved motor function or reaction time than when no therapy was given around the stimulation. Several other review articles and studies suggest using both high definition tDCS, which increases the focality of the current, and/or using neurotargeting software that uses the patient's own CT/MRI in the computation of the electrical montage can create a more personalized tDCS regimen.7,11,12 This study plans to do both. The Soterix MxN neuromodulation system has been used in multiple studies and has a targeting system that would help ensure both ideal current, more focal stimulation and optimal lead placements is essential as according to Datta et al (2011). Lesions within the brain may alter the flow of current through that area. The software system, HD-Targets, will be used that takes the patient's own MRI to account for variabilities in skull thickness, lesion size/location/composition, fluid density, and cerebrospinal fluid presence. These variabilities are used in the computer algorithm that simulates current flow through that specific participant's brain to get to the desired target area with the least amount of current and decreased stimulation of undesired areas. The investigators will examine these patients before and after treatment and compare the two groups, treatment group and sham group, after they receive 10 sessions of 20minutes along with their regular course of physical, occupational, or speech therapy over the course of their inpatient rehab stay.

Subjects will be given high definition transcranial direct current stimulation (tDCS) via a Soterix MxN HD-tDCS stimulator. This device is for investigational use only at this time and is not FDA approved. However, it has been used in several multicenter and randomized control trials that are detailed below in Appendix 1. The patient's MRi will be sent out to Soterix where they will manually input the variations in skull thickness, fluid density, lesion size, cerebrospinal fluid, and gray/white matter variabilities. They will then run the algorithm with HD-Targets, sophisticated current simulating software, to obtain optimal electrode placement to target the primary motor cortex (M1 area), the region of the brain that is responsible for movement, of each individual patient. Another issue with tDCs is maintaining optimal connections between the patient's scalp and the electrodes. Sotetrix HD-tDCs uses SmartScan™ to assure proper lead contact with initial set-up to adjust electrodes and head-gear for optimal fit. During stimulation, SmartScan™ provides a constant indication of electrode quality and can be monitored during adjustments to assure continuous lead contact.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18-90 years old
2. Diagnosed with middle cerebral artery ischemic stroke
3. Upper extremity movement deficits
4. Cardiorespiratory function is stable
5. Admitted to acute inpatient rehabilitation
6. Intact corticospinal tract

Exclusion Criteria:

1. Previous stroke
2. Pre-stoke weakness or disability in the paretic arm
3. Severe neglect
4. Acute exacerbation of heart failure or COPD
5. Severe aphasia
6. Decisional Impairment
7. Pregnant or nursing women
8. Prisoner
9. Skin disorder or wound of scalp
10. Seizure disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-05 (Estimated); Primary Completion 2022-09-05 (Estimated); Study Completion 2022-09-05 (Estimated)

PRIMARY OUTCOMES:
Change in the Fugl-Meyer upper extremity assessment | Assessments will be taken at baseline and after treatment (about 2 weeks) to determine change in the score after the treatments or sham stimulation has been given.
  It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It measures performances on motor function of the upper extremity. Range is from 0-66 with 66 being totally normal in all assessments. Each Sub score for each category ranges from 0-2 with 0 being not able to finish and 2 meaning function is normal in this category.

SECONDARY OUTCOMES:
Change in the Wolf Motor Function Test | Assessments will be taken at baseline and after treatment (about 2 weeks) to determine change in the score after the treatments or sham stimulation has been given.
  Quantifies upper extremity (UE) motor ability through timed and functional tasks. Thus, it measures how well a task can be performed by the subject, and the patient is given a score from 0-6. Zero being did not perform, and six being normal. The changes in performance can be compared over time to assess their progress. Each task is subscaled from 0-6 with 6 being indepednetly performed and 0 being unable to perform or needs to be performed by someone else for the patient.
Change in the Functional Independence Measure | Assessments will be taken at baseline and after treatment (about 2 weeks) to determine change in the score after the treatments or sham stimulation has been given.
  A uniform system of measurement for disability based on the International Classification of Impairment, Disabilities and Handicaps for use in the medical system in the United States. It is a measure of a person's physical, psychological, and social functions to assess their level of disability. It is a scale from 18-126 with a score of 126 being completely normal or independent in all of the tasks. 17 tasks in total: 6 are functional tasks, 2 measure strength, and 9 analyze movement quality or efficiency. Each task is subscored from 1-7 with 7 being completely independent completing a task and 1 meaning the person is fully dependent on someone completing that task for them.
Change in the Action Research Arm Test | Assessments will be taken at baseline and after treatment (about 2 weeks) to determine change in the score after the treatments or sham stimulation has been given.
  Evaluative measure to assess specific changes in limb function among individuals who sustained cortical damage resulting in hemiplegia (Lyle, 1981). This measures 19 items covering four domains of upper extremity movement: grasp, grip, pinch, and gross motor. Score ranges from 0-57 with 57 being normal function in all domains. Each task has a subscore of 0-3 with 0 being unable to perform movement and 3 being normal function.
Kinematic measurements with Kinereach system: measurement of change arm speed | Assessments will be taken at baseline and after treatment (about 2 weeks) to determine change in the score after the treatments or sham stimulation has been given.
  Developed by Robert Sainburg. The machine is able to measure how fast a patient's arm is able to move through space. Speed would be quantified as the peak and/or average tangential velocity of the hand during self-paced reaching movements.
Kinematic measurements with Kinereach system: measurement of change in arm smoothness | Assessments will be taken at baseline and after treatment (about 2 weeks) to determine change in the score after the treatments or sham stimulation has been given.
  Developed by Robert Sainburg. The machine is able to measure how smooth a patient is able to move their arm through space. Smoothness is measured as mean squared Jerk: This is quantified as the third derivative of displacement (jerk) squared and averaged over time.
Kinematic measurements with Kinereach system: measurement of change in arm range of motion | Assessments will be taken at baseline and after treatment (about 2 weeks) to determine change in the score after the treatments or sham stimulation has been given.
  Developed by Robert Sainburg. The machine is able to measure range of motion that would be quantified as the largest 2D area encircled by the hand, when asked to make the biggest circle possible. .
Change in National institute of Health Stroke Scale | Assessments will be taken at baseline and after treatment (about 2 weeks) to determine change in the score after the treatments or sham stimulation has been given.
  15-item impairment scale, intended to evaluate neurologic outcome and degree of recovery for patients with stroke. Range of scores from 0-42 with zero being no symptoms and 42 being severely impaired. It is a way to quantify stroke severity with measures for the typical stroke symptoms including level on consciousness, language, vision, motor and sensory involvement, as well as some cognitive assessments.
Change in Modified Rankin Scale | Assessments will be taken at baseline and after treatment (about 2 weeks) to determine change in the score after the treatments or sham stimulation has been given.
  Single item, global outcomes rating scale for patients post-stroke. Range is from 0-6. Zero being no symptoms and 6 being dead. In-between measures consist of how much help they require during their activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: William A Pomilla, MD, Principal Investigator — Assistant Professor

IPD SHARING:
Plan to Share IPD: No
No identifying data will be distributed. Demographic information with used within the groups to assess treatment versus sham homogenicity

REFERENCES:
- [Background] Di Pino G, Pellegrino G, Assenza G, Capone F, Ferreri F, Formica D, Ranieri F, Tombini M, Ziemann U, Rothwell JC, Di Lazzaro V. Modulation of brain plasticity in stroke: a novel model for neurorehabilitation. Nat Rev Neurol. 2014 Oct;10(10):597-608. doi: 10.1038/nrneurol.2014.162. Epub 2014 Sep 9. PMID 25201238
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. Neuroscientist. 2011 Feb;17(1):37-53. doi: 10.1177/1073858410386614. PMID 21343407
- [Background] Nitsche MA, Fricke K, Henschke U, Schlitterlau A, Liebetanz D, Lang N, Henning S, Tergau F, Paulus W. Pharmacological modulation of cortical excitability shifts induced by transcranial direct current stimulation in humans. J Physiol. 2003 Nov 15;553(Pt 1):293-301. doi: 10.1113/jphysiol.2003.049916. Epub 2003 Aug 29. PMID 12949224
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Elsner B, Kwakkel G, Kugler J, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving capacity in activities and arm function after stroke: a network meta-analysis of randomised controlled trials. J Neuroeng Rehabil. 2017 Sep 13;14(1):95. doi: 10.1186/s12984-017-0301-7. PMID 28903772
- [Background] Giordano J, Bikson M, Kappenman ES, Clark VP, Coslett HB, Hamblin MR, Hamilton R, Jankord R, Kozumbo WJ, McKinley RA, Nitsche MA, Reilly JP, Richardson J, Wurzman R, Calabrese E. Mechanisms and Effects of Transcranial Direct Current Stimulation. Dose Response. 2017 Feb 9;15(1):1559325816685467. doi: 10.1177/1559325816685467. eCollection 2017 Jan-Mar. PMID 28210202
- [Background] Rabadi MH, Aston CE. Effect of Transcranial Direct Current Stimulation on Severely Affected Arm-Hand Motor Function in Patients After an Acute Ischemic Stroke: A Pilot Randomized Control Trial. Am J Phys Med Rehabil. 2017 Oct;96(10 Suppl 1):S178-S184. doi: 10.1097/PHM.0000000000000823. PMID 28837443
- [Background] Kang N, Summers JJ, Cauraugh JH. Transcranial direct current stimulation facilitates motor learning post-stroke: a systematic review and meta-analysis. J Neurol Neurosurg Psychiatry. 2016 Apr;87(4):345-55. doi: 10.1136/jnnp-2015-311242. Epub 2015 Aug 28. PMID 26319437
- [Background] Hummel FC, Celnik P, Pascual-Leone A, Fregni F, Byblow WD, Buetefisch CM, Rothwell J, Cohen LG, Gerloff C. Controversy: Noninvasive and invasive cortical stimulation show efficacy in treating stroke patients. Brain Stimul. 2008 Oct;1(4):370-82. doi: 10.1016/j.brs.2008.09.003. Epub 2008 Oct 9. PMID 20633395
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Woods AJ, Antal A, Bikson M, Boggio PS, Brunoni AR, Celnik P, Cohen LG, Fregni F, Herrmann CS, Kappenman ES, Knotkova H, Liebetanz D, Miniussi C, Miranda PC, Paulus W, Priori A, Reato D, Stagg C, Wenderoth N, Nitsche MA. A technical guide to tDCS, and related non-invasive brain stimulation tools. Clin Neurophysiol. 2016 Feb;127(2):1031-1048. doi: 10.1016/j.clinph.2015.11.012. Epub 2015 Nov 22. PMID 26652115
- [Background] Nitsche MA, Grundey J, Liebetanz D, Lang N, Tergau F, Paulus W. Catecholaminergic consolidation of motor cortical neuroplasticity in humans. Cereb Cortex. 2004 Nov;14(11):1240-5. doi: 10.1093/cercor/bhh085. Epub 2004 May 13. PMID 15142961
- [Background] Monte-Silva K, Kuo MF, Thirugnanasambandam N, Liebetanz D, Paulus W, Nitsche MA. Dose-dependent inverted U-shaped effect of dopamine (D2-like) receptor activation on focal and nonfocal plasticity in humans. J Neurosci. 2009 May 13;29(19):6124-31. doi: 10.1523/JNEUROSCI.0728-09.2009. PMID 19439590
- [Background] Kuo MF, Unger M, Liebetanz D, Lang N, Tergau F, Paulus W, Nitsche MA. Limited impact of homeostatic plasticity on motor learning in humans. Neuropsychologia. 2008;46(8):2122-8. doi: 10.1016/j.neuropsychologia.2008.02.023. Epub 2008 Feb 29. PMID 18394661
- [Background] Nitsche MA, Doemkes S, Karakose T, Antal A, Liebetanz D, Lang N, Tergau F, Paulus W. Shaping the effects of transcranial direct current stimulation of the human motor cortex. J Neurophysiol. 2007 Apr;97(4):3109-17. doi: 10.1152/jn.01312.2006. Epub 2007 Jan 24. PMID 17251360
- [Background] Kuo MF, Paulus W, Nitsche MA. Boosting focally-induced brain plasticity by dopamine. Cereb Cortex. 2008 Mar;18(3):648-51. doi: 10.1093/cercor/bhm098. Epub 2007 Jun 24. PMID 17591596
- [Background] Fregni F, Thome-Souza S, Nitsche MA, Freedman SD, Valente KD, Pascual-Leone A. A controlled clinical trial of cathodal DC polarization in patients with refractory epilepsy. Epilepsia. 2006 Feb;47(2):335-42. doi: 10.1111/j.1528-1167.2006.00426.x. PMID 16499758
- [Background] Ward NS, Newton JM, Swayne OB, Lee L, Thompson AJ, Greenwood RJ, Rothwell JC, Frackowiak RS. Motor system activation after subcortical stroke depends on corticospinal system integrity. Brain. 2006 Mar;129(Pt 3):809-19. doi: 10.1093/brain/awl002. Epub 2006 Jan 18. PMID 16421171
- [Background] Santisteban L, Teremetz M, Bleton JP, Baron JC, Maier MA, Lindberg PG. Upper Limb Outcome Measures Used in Stroke Rehabilitation Studies: A Systematic Literature Review. PLoS One. 2016 May 6;11(5):e0154792. doi: 10.1371/journal.pone.0154792. eCollection 2016. PMID 27152853
- [Background] Lin JH, Hsueh IP, Sheu CF, Hsieh CL. Psychometric properties of the sensory scale of the Fugl-Meyer Assessment in stroke patients. Clin Rehabil. 2004 Jun;18(4):391-7. doi: 10.1191/0269215504cr737oa. PMID 15180122
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386